CLINICAL TRIAL: NCT01251185
Title: Extracorporeal Shockwave Myocardial Revascularization(ESMR)Therapy For The Treatment of Chronic Heart Failure.
Brief Title: Extracorporeal Shockwave Myocardial Revascularization (ESMR) Therapy For The Treatment of Chronic Heart Failure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medispec (Industry)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESMR CHF-IL
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Congestive Heart Failure
Keywords: Extracorporeal Shockwave Therapy; Heart Failure; Congestive Heart Failure; Non-invasive; Device Trial; NYHA (New York Heart Association); Ischemic cardiomyopathy; Ischemia; Myocardial contractility
MeSH Terms: conditions — Heart Failure; Ischemia | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CHF (Experimental): Single-arm, open label, subjects with Congestive Heart Failure, with ischemic etiology.
  Interventions: Device: Cardiospec

INTERVENTIONS:
Device: Cardiospec — Non-invasive, low-intensity extracoporeal shockwaves at energy density of 0.99 mJ/mm2. 9 treatment sessions, 20 minutes each, over a period of 9 weeks (3 sessions on weeks 1, 5 and 9).
  Other Names: Cardiospec ESMR therapy; Extracorporeal Shockwave therapy; Extracorporeal myocardial Revascularization

SUMMARY:
Evaluation of non-invasive treatment modality, using low-intensity extracorporeal shockwaves for treatment of subjects diagnosed with Congestive Heart Failure, with ischemic etiology.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is male or female 18 years or older.
2. Patient is diagnosed with a Heart Failure with ischemic etiology. Diagnosis is based on medical history, complete physical evaluation, and echocardiography.
3. Patient has documented myocardial segments with impaired contractility. Diagnosis is based on Rest Echo.
4. Patient is diagnosed with no more than 50% of segments akinetic or dyskinetic Diagnosis is based on echocardiography.
5. Patient is classified as NYHA II to IV.
6. Patient should be on a stable dosage of medication for at least 6 weeks prior to enrollment.
7. Patients Ejection Fraction < 50%.
8. Patient is stable and without clinical events for > 3 months.
9. Patient has signed an informed consent form.
10. Patient's condition should be stable and should have a life expectancy of >12 months.
11. Patient's current and past medical condition and status will be assessed using previous medical history, physical evaluation, and the physicians (principle investigator's)medical opinion.

Exclusion Criteria:

1. Patient with intraventricular thrombus.
2. Severe COPD (patients with an FEV1 less than .8 liters).
3. Patient has chronic lung disease including emphysema and pulmonary fibrosis.
4. Patient has active endocarditis, myocarditis or pericarditis.
5. Patient is simultaneously participating in another device or drug study, or has participated in any clinical trial involving an experimental device or drug, including other drugs or devices enhancing cardiac neovascularization or any ESWT machine for neovascularization of a competitor company within 3 months of entry into the study.
6. Patients who are unwilling or unable to cooperate with study procedure.
7. Patients who are unwilling to quit smoking during the study procedure (including screening phase).
8. Patients who are diagnosed with severe valvular disease (regurgitation or stenosis).
9. Patient is pregnant.
10. Patient with a malignancy in the area of treatment without complete remission within 5 years(lungs, thorax, ribs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The change in the number of myocardial segments that improve their contractility(at rest and at stress)at 6 months post baseline evaluations, evaluated by echocardiography. | 6 months
  An echo examination shall be used to evaluate myocardial contractility post treatments.

SECONDARY OUTCOMES:
6 Minutes Walk Test (6MWT) | 6 months
  Evaluation of 6MWT time from baseline to 6 months post baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Hilton Miller, Professor, Principal Investigator — Tel Aviv Souraski Center
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel